CLINICAL TRIAL: NCT01996007
Title: Cross-sectional Study to Establish the Point Prevalence of Serotype 19A Pneumococcal Nasopharyngeal Carriage of Fully Vaccinated Children Aged 13-48 Months Following Introduction of PCV13.
Brief Title: Understanding Pneumococcal Carriage and Disease
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: OVG 2013/05
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2015-11

CONDITIONS: Meningitis; Septicaemia; Pneumonia
Keywords: Pneumococcus; Carriage; Children; Parents; Immunogenicity; PCV13
MeSH Terms: conditions — Meningitis; Toxemia; Pneumonia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Bacteria grown from nasopharyngeal swabs Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Children: Pneumococcal nasopharyngeal carriage and immunogenicity in children aged 6-48 months who have previously received PCV13
- Parents: Pneumococcal nasopharyngeal carriage and immunogenicity in parents of children also participating in the study

SUMMARY:
Pneumococcus is a bacteria that causes disease of the respiratory tract (pneumonia and middle ear infections), blood poisoning, and meningitis. It is frequently carried by people in back of the throat without symptoms. Pneumococcal carriage in the Thames Valley region has been studied over the last 12 years with carriage rates having been shown to be reflective of disease potential and hence vaccine effect. During this time pneumococcal vaccines have been introduced into the routine immunisation schedules of this community. The PCV7 (A vaccine against 7 types of pneumococcus) vaccine has subsequently been noted to have had a significant impact in reducing vaccine serotype carriage and disease. Herd protection (indirect protection of unvaccinated individuals) has also been implicated with vaccine serotypes not being carried in parents of vaccinated children. The most common serotype carried since the introduction of PCV7 is 19A, which is included in the PCV13 vaccine (A vaccine against 13 types of pneumococcus). PCV13 has superseded PCV7 in the routine immunisation schedule, however its impact on carriage and disease in this community is yet to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Children

* Parent/guardian of participant is willing and able to give informed consent for participation in the study.
* In good health as determined by a brief medical history and/or clinical judgement of the investigator
* Have received three doses of PCV13 as per infant immunisation schedule (as confirmed by red book or through vaccination history and age). Vaccination history will be confirmed by the child's GP or CHCD. The visit and sampling may still proceed if the vaccination history has not been confirmed beforehand and the participant subsequently excluded if they are found to not have received all three doses of PCV13.Aged 6-48 months and at least 28 days since their third PCV13 vaccination.
* Able (in the Investigators opinion) and willing to comply with all study requirements.

Parents/ Legal guardians

* Participant is willing and able to give informed consent for participation in the study.
* Is the child's legal guardian and lives in the same household with the child participating in the same study.
* In good health as determined by clinical judgement of the research staff
* Able (in the investigators opinion) and willing to comply with all study requirements.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

Children

* Parent/legal guardian unwilling or unable to give written informed consent to participate in the study.
* Parent/legal guardian less than 18 years of age at time of enrolment.
* Parent/legal guardian is listed on the study delegation log.
* Children who are unimmunised or have an incomplete course of PCV13.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Febrile illness or temperature of 38°C on the day of the visit or in the preceding 24 hours.
* Respiratory illness on the day of the study visit or in the preceding 24 hours. A respiratory illness will be classified as a combination of at least two of the following symptoms: cough, sore throat, and runny nose.
* Administration of antibiotics in the month prior to sampling.
* A risk of nose bleed, including; a recent (within the last 24 hours) nose bleed, history of a bleeding disorder, history of severe nose bleeds or recent (within the last 3 months) nasal/craniofacial surgery.
* Receipt of blood products and/or plasma derivatives or any parenteral immunoglobulin preparation within 90 days.

Parents/ Legal guardians

* Participants who are unwilling or unable to give written informed consent to participate in the study.
* Less than 18 years of age at time of enrolment
* Is listed on the study delegation log
* Previous immunisation with pneumococcal conjugate vaccine.
* Participants who in the opinion of the investigator are unable to comply with study procedures or may be put at risk by participation in the study.
* Febrile illness or temperature of 38°C on the day of the visit or in the preceding 24 hours.
* Respiratory illness on the day of the study visit or in the preceding 24 hours. A respiratory illness will be classified as a combination of at least two of the following symptoms: cough, sore throat, and runny nose.
* Administration of antibiotics in the month prior to sampling.
* A risk of nose bleed, including; a recent (within the last 24 hours) nose bleed, history of a bleeding disorder, a history of severe nose bleeds or recent (within the last 3 months) nasal/craniofacial surgery.
* Receipt of blood products and/or plasma derivatives or any parenteral immunoglobulin preparation within 90 days.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: One thousand healthy children aged 6-48 months, of which at least 600 will be aged 21-48 months, who have received 3 doses of PCV13 will be recruited along with a subset (200) of their parents/legal guardians
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The presence of serotype 19A pneumococci on children's swabs | 2 years

SECONDARY OUTCOMES:
The presence of pneumococcal serotypes on children's swabs | 2 years
The presence of pneumococcal serotypes on parents/legal guardians swabs | 2 years
The molecular sequence type of nasopharyngeal carriage isolates from children and parents/legal guardians. | 2 years
The serotype-specific and genotype-specific invasive disease potential of isolates recovered from children. | 2 years
The serotype specific pneumococcal antibodies levels in children and their parents/legal guardians | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Pollard, PhD, Principal Investigator — Oxford Vaccine Group
Locations (1):
- Oxford Vaccine Group, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Result] Kandasamy R, Voysey M, Collins S, Berbers G, Robinson H, Noel I, Hughes H, Ndimah S, Gould K, Fry N, Sheppard C, Ladhani S, Snape MD, Hinds J, Pollard AJ. Persistent Circulation of Vaccine Serotypes and Serotype Replacement After 5 Years of Infant Immunization With 13-Valent Pneumococcal Conjugate Vaccine in the United Kingdom. J Infect Dis. 2020 Mar 28;221(8):1361-1370. doi: 10.1093/infdis/jiz178. PMID 31004136